CLINICAL TRIAL: NCT05136560
Title: A Randomized, Double-blind, Multi-center Clinical Trial to Evaluate the Safety and Efficacy of Early Administration of Dexamethasone in High-risk Sepsis
Brief Title: Safety and Efficacy of Early Administration of Dexamethasone in High-risk Sepsis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CHA University (Other)
Responsible Party: Principal Investigator, Kyuseok Kim, Professor, Emergency Department, CHA University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DEXA-SEPSIS
Record Dates: First submitted 2021-11-15; First posted 2021-11-29 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Sepsis
Keywords: sepsis, glucocorticoid
MeSH Terms: conditions — Sepsis | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (No Intervention): normal saline
- low dose dexamethasone (Experimental): 0.1 mg/kg dexamethasone iv once per day, for 1 or 2 days
  Interventions: Drug: Dexamethasone
- high dose dexamethasone (Experimental): 0.2 mg/kg dexamethasone iv once per day, for 1 or 2 days
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Intervention drugs would be administered for 1 or 2 days.
  Other Names: JEIL Dexamethasone Injection
  Arms: high dose dexamethasone; low dose dexamethasone

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of early administration of two different doses of dexamethasone in high risk septic patients.

DETAILED DESCRIPTION:
The septic adult patients of high risk would be enrolled in 2 emergency departments.

Sepsis would be defined by Sepsis-3 definition. High risk is defined as initial systolic blood pressure less than 90 mmHg or blood lactate level over 2 mmol/L.

The enrolled patients would be randomized to 3 groups: control, low dose dexamethasone (0.1 mg/kg iv), and high dose dexamethasone (0.2mg/kg iv).

The study drug is blinded and administered after enrollment for 2 days. Sample size would be 102, considering 10% of drop-out rate, allocating 30 patients to each groups.

Efficacy would be evaluated as follows; 28 day and 90 day mortality, time to septic shock, time to shock reversal, administration of steroid according to guideline, ventilator free days, Continuous renal replacement, Length of stay in ICU or hospital, delta SOFA score on day 3 and day 7,

Safety would be evaluated as follows; Superinfection Gastrointestinal bleeding, Hyperglycemia, Hypernatremia

ELIGIBILITY:
Inclusion Criteria:

* Sepsis defined by Sepsis-3 definition
* Initial systolic blood pressure < 90mmHg or blood lactate level >2mmol/L

Exclusion Criteria:

* advanced directive for "Do not resuscitation"
* recent systemic administration of glucocorticoid (4 weeks)
* recent systemic administration of chemotherapy (4 weeks)
* recent systemic administration of immunosuppressant (4 weeks)
* expected life less than 90 days
* Transferred from other hospital
* Sepsis diagnosed 24 hours after ED admission
* Use of etomidate in ED
* pregnant or on lactation
* no informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
28 day mortality | 28 days
  death at 28 day

SECONDARY OUTCOMES:
90 day mortality | 90 days
  death at 90 day
Time to septic shock | up to 1 month, During hospital stay
  Time to septic shock after enrollment
Time to shock reversal | up to 1 month, During hospital stay
  time required for shock reversal
Administration of steroid according to guideline, yes or no | up to 1 month, During hospital stay
  Need for additional steroid requirement according to the sepsis guideline
ventilator free days | up to 3 month, During hospital stay
  days independent from ventilator care
continuous renal replacement therapy (CRRT) | up to 3 month, During hospital stay
  requirement of CRRT
Length of stay in intensive care unit (ICU) | up to 6 month, During hospital stay
  Days spent in intensive care unit (ICU)
Length of stay in hospital | up to 6 month, During hospital stay
  Days spent in hospital
Delta SOFA sore on day 3 and 7 | 7 days
  Change of SOFA score on day 3 and day 7
Superinfection | 28 days
  secondary infection
Gastrointestinal bleeding | 14 days
  Gastrointestinal bleeding at any amount
Hyperglycemia | 7 days
  serum glucose >150 mg/dL
Hypernatremia | 7 days
  serum sodium >150mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Kyuseok Kim, M.D, PhD, Principal Investigator — Bundang CHA Hospital
Locations (2):
- South Korea (2):
  - Bundang CHA hospital, Seongnam-si, Gyeonggi-do
  - Samsung Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Choi K, Park JE, Kim A, Hwang S, Bae J, Shin TG, Kim K. The DEXA-SEPSIS study protocol: a phase II randomized double-blinded controlled trial of the effect of early dexamethasone in high-risk sepsis patients. Clin Exp Emerg Med. 2022 Sep;9(3):246-252. doi: 10.15441/ceem.22.276. Epub 2022 Sep 20. PMID 36116775